CLINICAL TRIAL: NCT02379624
Title: Pectin Start Early Enteral Nutritional Support in Critically Ill Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xingwei Xu (Other)
Responsible Party: Sponsor-Investigator, Xingwei Xu, Doctor, Nanjing University
Organization: Nanjing University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NNSF81270884
Record Dates: First submitted 2014-08-30; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Nutrition Disorders; Critical Illness
MeSH Terms: conditions — Nutrition Disorders; Critical Illness | interventions — Pectins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EN group (Placebo Comparator): 5% glucose at a rate of 25 mL/h was given at day 1, followed with initial amount of EN (31.25g peptisorb dissolved in 250ml water) at 12.5 mL/h on day 2. From day 3 to day 6, the prescription is EN (62.5g peptisorb dissolved in 250ml water) at 12.5 mL/h. Since day 7, EN was began to advance to goal energy target as quickly as possibl
- PEC/EN group (Experimental): An additional amount of pectin was added 4 hours ahead of EN given from day 2 to day 6 (24g everday). Since day 7, EN was advanced to goal energy target as the same step
  Interventions: Drug: pectin

INTERVENTIONS:
Drug: pectin — Pectin, a representative diety fibre, is a gelatinous substance derived from the cell walls of fruits and some plants and contains galacturonan, consisting of mostly long-chain D-galacturonic acids combined into units by α-1,4 linkages. As a kind of soluble dietary fiber, pectin has been proved of controlling glucose and blood lipids. It slows rapid infusion of the liquid meal into the gut by delaying gastric emptying.
  Arms: PEC/EN group

SUMMARY:
Acute lower gastrointestinal dysfunction is a kind of much common complication which occurred in critically ill patients. Once it developed, enteral nutrition would be disturbed. In this study, investigators suppose that early application of a sufficient amount of pectin ahead of enteral nutrition, may promote recovery of acute lower gastrointestinal dysfunction in critically ill patients, and exert its good effect on early EN support.

Investigators designed this prospective randomized controlled trial to test and evaluates the effect whether EN feeding with or without a pectin start would be safe or with advanced clinical outcomes.

DETAILED DESCRIPTION:
Gastrointestinal function (GI) is an important determinant in the outcome of critically ill patients, with up to 62% of patients exhibiting at least one GI symptom for at least 1 day. Unlike the upper gastrointestinal dysfunction, which can be diagnosed early because of abdominal distension, nausea, and feeding intolerance, acute lower gastrointestinal dysfunction (ALGID) is a kind of more common complication which more easily neglected due to atypical symptoms. Once ALGID developed, critical patients could not get enteral nutrition (EN) normally, as early EN support is often essential and standard on critically ill patients when feasible. It also causes colonic bacteria reflux to the ileum and jejunum, leads to ischemic necrosis or colon perforation, and increases the incidence of various adverse events.

Dietary fiber (DF) plays an important and helpful role in GI. It undergoes partial or total fermentation in the distal small bowel and colon, leading to the production of short chain fatty acids (SCFA) and gas. It also helps to conduct slower and delayed gastroenterology absorption, and reduce luminal flow. To date, many research and evidences exist for DF-supplemented EN reduces the incidence of colonic dysfunction in non-intensive care unit studies. However, until recently, it still lacks guidelines on how to conduct DF-supplemented EN rationally in critically ill patients.

Pectin, a representative DF, is a gelatinous substance derived from the cell walls of fruits and some plants and contains galacturonan, consisting of mostly long-chain D-galacturonic acids combined into units by α-1,4 linkages. As a kind of soluble dietary fiber, pectin has been proved of controlling glucose and blood lipids. It slows rapid infusion of the liquid meal into the gut by delaying gastric emptying. Studies showed that 90% of ingested pectin can be found in the terminal ileum. In view of all the former studies data and on the basis of investigators' clinical observation, investigators postulate that early application of a sufficient amount of pectin ahead of EN, may promote ALGID recovery in critically ill patients, and exert its effect.

Investigators designed this prospective randomized controlled trial to test whether EN feeding with or without a pectin start would be safe or with advanced clinical outcomes. Investigators speculated that pectin start EN could nourish the digestive tract in critically ill patients, and it is superior to traditional EN feeding for the delivery of early nutritional support.

ELIGIBILITY:
Inclusion Criteria:：

* Adult ICU patients who were at least 18 years old if they were expected to require EN support within 36 hours after an unplanned ICU admission.

Exclusion Criteria:

* Could not be fed through enteral route,
* Had received EN in the past 2 months,
* Had a colectomy or jejunostomy in situ,
* Had severe colonic disease such as ulcerative colitis and Crohn's,
* Had pregnant,
* Had EN taboo crowd.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2014-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | 30 days

SECONDARY OUTCOMES:
duration of organ support | 30 days
Efficacy as measured by frequency of treated infectious and noninfectious complications | 30 days
Efficacy as measured by frequency of Vomiting | 30 days
Efficacy as measured by frequency of Diarrhea | 30 days
Efficacy as measured by frequency of Abdominal distention or Cramping | 30 days
Efficacy as measured by frequency of Constipation | 30 days
Efficacy as measured by frequency of Regurgitation | 30 days
Efficacy as measured by frequency of Given antidiarrheal | 30 days
Efficacy as measured by frequency of Given prokinetic agents | 30 days